CLINICAL TRIAL: NCT06884488
Title: Effect of Preconditioning of Human Pharyngeal Motor Cortex by Low Frequency Repetitive Transcranial Magnetic Stimulation on Enhancing Cortical Excitability Induced by Pharyngeal Electrical Stimulation
Brief Title: Aftereffects of PES Preconditioned with RTMS on the Human Pharyngeal Motor Cortex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Prof Shaheen Hamdy PhD FRCP, Professor, University of Manchester
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-20990-37010
Record Dates: First submitted 2025-02-27; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Subjects (HS)
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- real rTMS + real PES (Experimental): Participants will receive real 1Hz rTMS over the dominant hemisphere, followed by a 30min interval. After that the participants will receive real 5Hz PES.
  Interventions: Device: repetitive transcranial magnetic stimulation (Magstim Super Rapid stimulator, The Magstim Company Ltd, Whitland, UK); Device: pharyngeal electrical stimulation (Digitimer model DS7; Welwyn-Garden City, Herts, UK)
- sham rTMS + real PES (Sham Comparator): Participants will receive sham 1Hz rTMS over the dominant hemisphere, followed by a 30min interval. After that the participants will receive real 5Hz PES.
  Interventions: Device: pharyngeal electrical stimulation (Digitimer model DS7; Welwyn-Garden City, Herts, UK); Device: sham repetitive transcranial magnetic stimulation(Magstim Super Rapid stimulator, The Magstim Company Ltd, Whitland, UK)
- real rTMS + sham PES (Sham Comparator): Participants will receive real 1Hz rTMS over the dominant hemisphere, followed by a 30min interval. After that the participants will receive sham 5Hz PES.
  Interventions: Device: repetitive transcranial magnetic stimulation (Magstim Super Rapid stimulator, The Magstim Company Ltd, Whitland, UK); Device: sham pharyngeal electrical stimulation (Digitimer model DS7; Welwyn-Garden City, Herts, UK)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (Magstim Super Rapid stimulator, The Magstim Company Ltd, Whitland, UK) — The paradigm will be applied over the dominant cerebral hemisphere for 10 minutes (600 pulses) over the dominant pharyngeal motor cortex capped at 120% of pharyngeal resting motor threshold.
  Arms: real rTMS + real PES; real rTMS + sham PES
Device: pharyngeal electrical stimulation (Digitimer model DS7; Welwyn-Garden City, Herts, UK) — The PES (0.2-ms pulses, 280 V) was delivered at a set frequency (5 Hz), intensity (75% of maximal tolerated), and duration (10 minutes), which have been reported as the most effective parameters for PES.
  Arms: real rTMS + real PES; sham rTMS + real PES
Device: sham repetitive transcranial magnetic stimulation(Magstim Super Rapid stimulator, The Magstim Company Ltd, Whitland, UK) — Sham rTMS is delivered with the coil tilted to its side at 90 degrees and with the identical stimulation conditions as active 1 Hz rTMS.
  Arms: sham rTMS + real PES
Device: sham pharyngeal electrical stimulation (Digitimer model DS7; Welwyn-Garden City, Herts, UK) — For sham pharyngeal stimulation, the same method including the insertion of the catherter will be employed without actual electrical stimulation.
  Arms: real rTMS + sham PES

SUMMARY:
The goal of this interventional study is to optimize the excitatory brain effects of combined neuromodulatory therapies on swallowing areas of the brain. The main question it aims to answer is:

Does preconditioning with 1 Hertz (Hz) repetitive transcranial magnetic stimulation (rTMS) delivered over hemispheric pharyngeal areas enhance the activating effects of pharyngeal electrical stimulation (PES) on cortical excitability?

Participants will:

* Visit the department three times, with at least a one-week gap between visits.
* Undergo baseline measurements for Pharyngeal motor evoked potential (PMEP) and Thenar motor evoked potential (TMEP), involving an electromyography (EMG) pharyngeal catheter inserted into the pharynx and gel electrodes to detect muscle activity.
* Be randomly allocated to one of the three preconditioning-conditioning procedures during each visit : 1Hz rTMS followed by 5Hz PES, sham 1Hz rTMS followed by 5Hz PES, and 1Hz rTMS followed by sham 5Hz PES

  1. Real rTMS will involve a figure-of-eight coil flat against the head delivering 1Hz stimulation at 90% of the thenar resting motor threshold.
  2. Sham rTMS will involve holding the coil perpendicular to the scalp to prevent brain stimulation.
  3. PES will involve a catheter delivering 0.2-ms pulses at 5Hz and 75% of the maximal tolerated intensity for 10 minutes. Sham PES will involve deactivating the current generator.
* Complete PMEP and TMEP measurements at baseline before intervention and every 15 minutes from 0 - 60 minutes after the rTMS-PES procedure.
* Complete a survey regarding tolerability and safety at the end of each visit.

DETAILED DESCRIPTION:
1 Study design This is a cross-over study with the order of experimental conditions randomized for each participant. The randomisation will be conducted using a randomisation program (Stats Direct, v2.7.8, StatsDirect Ltd, Altrincham, UK). Each condition will be given on separate days, at least one week apart.

2. Participants Healthy volunteers over the age of 18 will be recruited through adverts placed around Salford Royal Hospital, on a University of Manchester website which advertises for research volunteers and through a departmental database of volunteers who have expressed an interest in future research.

3. Informed consent A participant information sheet will be given to each participant. A researcher with up-to-date Good Clinical Practice (GCP) training will be responsible for obtaining consent from the participants. He/she will explain the study purpose and nature and experimental procedures verbally to the participants. The participants will be given sufficient time (at least 24 hours) to read and digest the written information and discuss with the researcher about the study. The researcher will ensure the participants are volunteering to participate, understand the purpose and nature, experimental procedures, benefits and risks of the study before obtaining written consent from them. The participants should understand that they have the rights to withdraw from the study anytime throughout the study.

4. Study Procedures

Participants will undergo either active or sham preconditioned 1 Hz rTMS interventions with 30 min intervals before active or sham 5 Hz PES (Fig 1). Each session involved:

1. A baseline measurement of PMEP and TMEP.
2. Application of (active/sham) 1 Hz rTMS (preconditioning).
3. A resting interval (30 minutes).
4. Application of (active/sham) 5 Hz PES (conditioning).
5. Measurement of PMEP and TMEP at multiple time points (immediately, 15, 30, 45, and 60 minutes post-PES).

5. End of study The study will come to an end after the period of data collection and analysis by the end of August 2025.

6. Withdraw consent Participants are able to withdraw consent at any time they wish. This will be stressed to all participants by members of the research team. Should this happen, their data will be retained with permission from the subject and they will be removed from the study.

As only healthy participants will be recruited for this study, no participant is expected to lose the capacity to consent during the course of the study. However, if for any reason a loss of capacity is suspected, the participant will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers over the age of 18 will be recruited through adverts placed around Salford Royal Hospital, on a University of Manchester website which advertises for research volunteers and through a departmental database of volunteers who have expressed an interest in future research. There is no upper age limit for potential participants.

Exclusion Criteria:

The presence or a history of:

1. Epilepsy
2. Cardiac pacemaker
3. Previous brain surgery
4. Previous swallowing problems
5. The use of medication which acts on the central nervous system
6. Any implanted metal in the head
7. Pregnancy (self-declared)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change of the amplitude of PMEP after intervention | Before intervention, 0 minutes, 15 minutes, 30 minutes, 45 minutes, and 60 minutes after the intervention
  The percentage change (in percents) of the amplitude (in millivolts) of bilateral PMEPs at different timepoints after the full intervention will be calculated as compared with the baseline measurement before the intervention.
Percentage change of the latency of PMEP after intervention | Before intervention, 0 minutes, 15 minutes, 30 minutes, 45 minutes, and 60 minutes after the intervention
  The percentage change (in percents) of the latency (in milliseconds) of bilateral PMEPs at different timepoints after the full intervention will be calculated as compared with the baseline measurement before the intervention.

SECONDARY OUTCOMES:
Percentage change of the amplitude of TMEP after intervention | Before intervention, 0 minutes, 15 minutes, 30 minutes, 45 minutes, and 60 minutes after the intervention
  The percentage change (in percents) of the amplitude (in millivolts) of bilateral TMEPs at different timepoints after the full intervention will be calculated as compared with the baseline measurement before the intervention.
Percentage change of the latency of TMEP after intervention | Before intervention, 0 minutes, 15 minutes, 30 minutes, 45 minutes, and 60 minutes after the intervention
  The percentage change (in percents) of the latency (in milliseconds) of bilateral TMEPs at different timepoints after the full intervention will be calculated as compared with the baseline measurement before the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Hamdy, PhD, Principal Investigator — The University of Manchester
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No